CLINICAL TRIAL: NCT00974753
Title: A Placebo-controlled, Randomized, Clinical Trial of Prophylactic Ketorolac 0.5% in Patients Undergoing Pars Plana Vitrectomy and Phacovitrectomy Epiretinal Membrane Peel Surgery: Assessing Macular Volume With Spectral-domain OCT
Brief Title: Prophylactic Ketorolac Post Epiretinal Membrane Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ERM-JG-2009
Record Dates: First submitted 2009-09-08; First posted 2009-09-10 (Estimated); Last update posted 2016-01-13 (Estimated); Status verified 2016-01

CONDITIONS: Macular Edema
Keywords: epiretinal membrane
MeSH Terms: conditions — Macular Edema; Epiretinal Membrane | interventions — Ketorolac Tromethamine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- PPV-MP + Placebo (Saline drops) (Placebo Comparator): PPV-MP= pars plana vitrectomy membrane peel
  Interventions: Other: Saline drops
- PPV-MP + Ketorolac 0.5% (Active Comparator): PPV-MP= pars plana vitrectomy membrane peel
  Interventions: Drug: Ketorolac 0.5%
- PhacoVit-MP + Placebo (Saline drops) (Placebo Comparator): PhacoVit-MP= phacovitrectomy membrane peel
  Interventions: Other: Saline drops
- PhacoVit-MP + Ketorolac 0.5%. (Active Comparator): PhacoVit-MP= phacovitrectomy membrane peel
  Interventions: Drug: Ketorolac 0.5%

INTERVENTIONS:
Drug: Ketorolac 0.5% — Four-times a day starting one week before surgery and continued for 4 weeks post surgery.
  Other Names: ketorolac tromethamine; Apo-Ketorolac
  Arms: PPV-MP + Ketorolac 0.5%; PhacoVit-MP + Ketorolac 0.5%.
Other: Saline drops — Four-times a day starting one week before surgery and continued for 4 weeks post surgery.
  Arms: PPV-MP + Placebo (Saline drops); PhacoVit-MP + Placebo (Saline drops)

SUMMARY:
Evaluate the efficacy of ketorolac 0.5%, a topical non-steroidal anti-inflammatory drug (NSAID), to prevent macular edema after epiretinal membrane surgery. Patients undergoing epiretinal membrane surgery have increased risk of macular swelling which can adversely affect vision. Since post-intraocular surgery inflammation is a contributing factor to macular swelling and loss of vision, NSAID drops may be able to prevent or minimize the deleterious effects of macular swelling after epiretinal membrane surgery.

ELIGIBILITY:
Inclusion Criteria:

* idiopathic epiretinal membrane diagnosis requiring membrane peel surgery

Exclusion Criteria:

* proliferative diabetic retinopathy
* sickle cell retinopathy
* radiation retinopathy
* choroidal folds
* hypersensitivity or allergy to NSAIDs
* wet macular degeneration
* branch retinal vein occlusion (BRVO)
* central retinal vein occlusion (CRVO)
* complicated membrane peel surgery

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2010-03; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Change in macular volume from baseline. | Before surgery, at 1 week, 1 month, and 1 year after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Gale, MD, FRCSC, Principal Investigator — Queen's University
Locations (1):
- Department of Ophthalmology, Hotel Dieu Hospital, Queen's University, Kingston, Ontario, Canada